CLINICAL TRIAL: NCT01628341
Title: French Observational Survey to Assess Hypoglycaemia in Insulin-treated Diabetic Patients
Acronym: DIALOG
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3988; U1111-1131-8540 (Other: WHO)
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with diabetes (type 1 and 2)
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: insulin — Patients will be asked to complete 2 self-assessment questionnaires

SUMMARY:
This non-interventional study is conducted in Europe. The study is both retrospective and prospective.

The purpose of the study is to assess the frequency of hypoglycaemia (low blood glucose) in insulin-treated patients with type 1 and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 Diabetes Mellitus
* Patients treated by insulin for at least 12 months
* Patients able to perform capillary self-monitoring plasma glucose (SMPG) measurements
* Patients able to complete the questionnaires
* Patients who have accepted to participate to the survey (signature of an information notice)

Exclusion Criteria:

* Patients with Type 2 Diabetes Mellitus not treated with insulin
* Females who are currently pregnant or lactating or who were pregnant during the previous year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 3811 patients with Type 1 or Type 2 diabetes are expected to be recruited. Patients will be asked to complete 2 self-assessment questionnaires, one retrospective and one prospective, to characterize severe hypoglycaemias during the last 12 months (retrospective questionnaire) and severe/non-severe hypoglycaemias during the coming month after inclusion (prospective questionnaire).
Sampling Method: Non-Probability Sample
Enrollment: 4424 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percentage of insulin-treated patients experiencing at least one hypoglycaemia (severe/non-severe) | During the one-month follow-up after inclusion in study

SECONDARY OUTCOMES:
Percentage of insulin-treated patients experiencing at least one severe hypoglycaemia | During the last 12 months before inclusion in study
Percentage of insulin-treated patients experiencing at least one severe hypoglycaemia | During the one-month follow-up after inclusion in study
Percentage of insulin-treated patients experiencing at least one non-severe symptomatic hypoglycaemia | During the one-month follow-up after inclusion in study
Percentage of insulin-treated patients experiencing at least one asymptomatic hypoglycaemia | During the one-month follow-up after inclusion in study
Percentage of insulin-treated patients experiencing at least one hypoglycaemia (overall/severe/non-severe) | During the one-month follow-up after inclusion in study
Rate of episodes (event/patient/month) in insulin-treated patients of severe hypoglycaemia | During the last 12 months before inclusion in study
Rate of episodes (event/patient/month) in insulin-treated patients of severe hypoglycaemia | During the one-month follow-up after inclusion in study
Rate of episodes (event/patient/month) in insulin-treated patients of non-severe symptomatic hypoglycaemia episodes | During the one-month follow-up after inclusion in study
Rate of episodes (event/patient/month) in insulin-treated patients of asymptomatic hypoglycaemia episodes | During the one-month follow-up after inclusion in study
Overall/severe/non-severe hypoglycaemia episodes (event/patient/month) | During the one-month follow-up after inclusion in study
Extra diagnostic tests carried out (number of extra self-monitoring plasma glucose (SMPG) test following the episode) | During the one-month follow-up after inclusion in study
Additional consultations to a specialist and/or general practitioner (GP), visit to emergency department, hospitalizations, transportation and assistance of a care-giver | During the one-month follow-up after inclusion in study
Change in planned daily activities; sleep, food consumption, physical activities (sport), driving, social life | During the one-month follow-up after inclusion in study
Change in planned daily activities; work: effectiveness, missing hours or days for sick leave | During the one-month follow-up after inclusion in study

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France

REFERENCES:
- [Result] Cariou B, Fontaine P, Eschwege E, Lievre M, Gouet D, Huet D, Madani S, Lavigne S, Charbonnel B. Frequency and predictors of confirmed hypoglycaemia in type 1 and insulin-treated type 2 diabetes mellitus patients in a real-life setting: results from the DIALOG study. Diabetes Metab. 2015 Apr;41(2):116-25. doi: 10.1016/j.diabet.2014.10.007. Epub 2014 Nov 24. PMID 25465273
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com